CLINICAL TRIAL: NCT03901079
Title: A Prospective, Multi-center, Non-Randomized Controled Trial for A Novel Facilitated Antegrade Steering Technique in Revascularization of Coronary Chronic Total Occlusions In Chinese Population--FAST CTO China
Brief Title: Trial for A Novel Facilitated Antegrade Steering Technique in Revascularization of Coronary Chronic Total Occlusions
Status: Terminated | Type: Observational
Why Stopped: HGRAC approval letter had expired. The enrollment speed of FAST CTO is much slower than planning and the scientific value becomes limited due to the delayed data readout anticipation.
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2362
Record Dates: First submitted 2018-08-10; First posted 2019-04-03 (Actual); Results first posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: CAD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CTO BridgePoint system: BridgePoint CTO System:
  * CrossBoss Catheter
  * Stingray LP Catheter
  * Stingray Guidewire and Extension Wire
  Interventions: Other: single-arm study

INTERVENTIONS:
Other: single-arm study — single-arm study

SUMMARY:
To assess the safety and efficacy of the BridgePoint CTO system in recanalization of CTO lesions which are resistant to a conventional wire approach in a multicenter study in Chinese population

DETAILED DESCRIPTION:
All subjects who are candidates for percutaneous coronary intervention (PCI), signed the informed consent form and had chronic total coronary occlusion (CTO) lesion will be evaluated for enrollment in this study.At least 100 subjects will be enrolled. Each site will be allowed to enroll up to a maximum of 25 subjects.

Primary Effectiveness Endpoint:

Technical Success: the ability of the BridgePoint Medical System to successfully facilitate placement of a guidewire beyond a CTO lesion in the true vessel lumen/within the collaterals in those cases that were otherwise refractory to treatment with a currently marketed guidewire

Primary Safety Endpoint:

30-day MACE rate for CTO cases in which the BridgePoint Medical System was used.

MACE is defined as the composite of cardiac death, Q-wave and non-Q-wave myocardial infarction(MI), and any ischemia-driven target lesion revascularization(TLR).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 but < 80 years of age
* Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed
* Subject is eligible for percutaneous coronary intervention (PCI)
* Subject has symptomatic coronary artery disease or myocardial infraction (MI) with objective evidence of ischemia or silent ischemia
* Subject is an acceptable candidate for coronary artery bypass grafting (CABG)
* Subject is willing to comply with all protocol-required follow-up evaluation
* Subject has a left ventricular ejection fraction (LVEF) ≥45% as measured within 60 days prior to enrollment

Angiographic Inclusion Criteria:

AI1. A maximum of one de novo CTO lesion in a native coronary artery with thrombolysis in Myocardial Infarction (TIMI) flow grade 0 AI2. Non-acute CTO lesion with an estimated duration of at least 3 months by clinical history and/or comparison with previous angiogram or electrocardiogram(ECG) AI3. The CTO lesion must have an angiographic landing zone≥ 10 mm proximal to any major bifurcation without severe calcification.

AI4. Lesion length < 40mm without excessive tortuosity and angulation(>45°)

Exclusion Criteria:

* Subject has clinical symptoms and/or ECG changes consistent with Acute MI (include STEMI and Non- STEMI) within 1 week
* Subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support, intractable ventricular arrhythmias, or ongoing intractable angina
* Subject has received an organ transplant or is on a waiting list for an organ transplant
* Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
* Planned PCI (including staged procedures) or CABG after the index procedure
* Subject has a known allergy to contrast (that cannot be adequately pre-medicated) and/or protocol-required concomitant medications (e.g., aspirin or all thienopyridines)
* Subject has one of the following (as assessed prior to the index procedure):

Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 12 months / Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.) / Planned procedure that may cause non-compliance with the protocol or confound data interpretation

* Subject is receiving chronic (≥72 hours) anticoagulation therapy (i.e., heparin, coumadin)
* Subject with out of range complete blood count (CBC) values that are determined by the study physician to be clinically significant.
* Subject is on dialysis or has baseline serum creatinine level >2.0 mg/dL (177µmol/L)
* Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Subject has had a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months
* Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding
* Subject has signs or symptoms of active heart failure (i.e., NYHA class IV) or LVEF < 45% at the time of the index procedure
* Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint or intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure
* Subject had PCI within the previous 2 weeks
* Subject with known intention to procreate within 12 months after the index procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure)
* Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)

Angiographic Exclusion Criteria:

AE1. Target lesion is an aorto-ostial lesion or located in left main coronary artery, previous venous or arterial bypass grafts AE2. Target lesion involving a segment of previous stent AE3. Target vessel has excessive tortuosity and/or angulation proximal to the target lesion(>45°) AE4. Target lesion and/or the target vessel proximal to the target lesion is moderately to severely calcified by visual estimate AE5. Target lesion is located within 5 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCx) coronary artery by visual estimate AE6. Target lesion will be accessed via a saphenous vein graft or arterial graft AE7. Subject has unprotected left main coronary artery disease (>50% diameter stenosis) AE8. Thrombus, or possible thrombus, present in the target vessel (by visual estimate) AE9. Target vessel has a dissection greater than National Heart, Lung, Blood Institute (NHLBI) type C

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who are candidates for percutaneous coronary intervention (PCI), signed the informed consent form and had chronic total coronary occlusion (CTO) lesion will be evaluated for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuejin Yang, Doc., Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- West China Hospital Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CTO BridgePoint System: BridgePoint CTO System:
  * CrossBoss Catheter
  * Stingray LP Catheter
  * Stingray Guidewire and Extension Wire
  single-arm study: single-arm study
Period: Overall Study
Arm/Group | CTO BridgePoint System
Started | 20 (There were 20 subjects enrolled totally.Due to the HGRAC approval letter expiration in August 2020 and cannot be extended on time，8 of the 20 subjects already enrolled were unable to complete the follow-up)
Completed | 12
Not Completed | 8
Not completed — 8 of the 20 subjects already enrolled were unable to complete the the 12-month follow-up | 8

BASELINE CHARACTERISTICS:
Population: Subject demographics, Physical assessment, Medical history, Angina assessment, LVEF, Cardiac medication, risk factors, and pre-procedure lesion characteristics will be summarized using descriptive statistics for continuous variables and frequency tables for discrete variables. No formal statistical testing will be done since this is a single-arm trial.
Arm/Group | CTO BridgePoint System
Number analyzed (Participants) | 20
Age, Continuous [Median (Standard Deviation); unit: years] | 57.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Current diabetes mellitus [Count of Participants; unit: Participants]
  Yes | 4
  No | 16
History of hyperlipidemia requiring medication [Count of Participants; unit: Participants]
  Yes | 18
  No | 2
History of hypertension requiring medication [Count of Participants; unit: Participants]
  Yes | 9
  No | 11
Family history of coronary artery disease [Count of Participants; unit: Participants]
  Yes | 3
  No | 16
  Unknown | 1
History of Myocardial Infarction (MI) [Count of Participants; unit: Participants]
  Yes | 3
  No | 17
History of congestive heart failure [Count of Participants; unit: Participants]
  Yes | 0
  No | 20
Current anginal status [Count of Participants; unit: Participants]
  None | 6
  Stable angina | 5
  Unstable angina | 8
  Unknown | 1
Does Subject have silent ischemia [Count of Participants; unit: Participants]
  Yes | 0
  No | 20
History of Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants]
  Yes | 8
  No | 12
History of Coronary Artery Bypass Graft (CABG) surgery [Count of Participants; unit: Participants]
  Yes | 0
  No | 19
  Unknown | 1
History of arrhythmia [Count of Participants; unit: Participants]
  Yes | 1
  No | 19
Left Ventricular Ejection Fraction (LVEF) measured [Count of Participants; unit: Participants]
  Yes | 19
  No | 1
History of cardiogenic shock [Count of Participants; unit: Participants]
  Yes | 0
  No | 20

OUTCOME MEASURES:

1. Primary Outcome: Technical Success: Successfully Facilitate Placement of a Guidewire Beyond a CTO Lesion in the True Vessel Lumen/Within the Collaterals
Description: 6 subjects have the results data, and 5 of them (83.3%) reported technical success. One (16.7%) failed.
Time Frame: Subject follow up will occur via telephone contact or clinic visit at 30 days,6 and 12 months post index procedure.
Population: Only 6 subjects have the results of technical success or not.
Measure: Count of Participants; unit: Participants
Arm/Group | CTO BridgePoint System
Number analyzed (Participants) | 6
Participants
  Success | 5
  Failed | 1

ADVERSE EVENTS:
Time Frame: Baseline,30 days, 6 months and 12 months
Arm/Group | CTO BridgePoint System
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CTO BridgePoint System (N=20)
Coronary artery atherosclerotic heart disease (Cardiac disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
HGRAC rejected all initiated applications from the leading site without any comments. Only leading site can submit the HGRAC application for multi-center studies and the ban lifting date of leading site is still unclear, it's not allowed to recruit or collect any data from the subjects after Aug 2020 (the expiry date of the approval ). The enrollment speed of FAST CTO is much slower than planning and the scientific value becomes limited due to the delayed data readout anticipation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT03901079/Prot_001.pdf
  • Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT03901079/SAP_002.pdf